CLINICAL TRIAL: NCT07030452
Title: Effectiveness and Safety of Laser Acupuncture on Pulmonary Function Test and Quality of Life in Patients With Chronic Obstructive Pulmonary Disease)
Brief Title: Laser Acupuncture for Pulmonary Function Test and Quality of Life in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dwi Lestari Ayuningtyas, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 25-05-0725
Record Dates: First submitted 2025-06-12; First posted 2025-06-22 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chronic Pulmonary Obstruction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The intervention group will receive laser acupuncture, while the control group will receive sham laser acupuncture
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be applied to participants and outcome assessor. Group allocation will not be disclosed to them to minimize assessment bias
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Laser Acupuncture
  Interventions: Device: Laser Acupuncture
- Control Group (Sham Comparator): Sham Laser Acupuncture
  Interventions: Device: Sham Laser Acupuncture

INTERVENTIONS:
Device: Laser Acupuncture — Laser acupuncture irradiation was performed using an RJ Laser laserpen with a wavelength of 785 nm and an output power of 50 mW. The laser probe was positioned perpendicularly to the skin surface, using a continuous wave mode with a dose of 4 Joules. The acupuncture points targeted were EXB1 and CV17, as well as BL13 and ST36 on both sides of the body. Each point received irradiation for 1 minute and 20 seconds. During the therapy session, subjects wore a headset playing music and protective glasses. The treatment was administered twice a week for a total of 8 sessions.
  Arms: Intervention Group
Device: Sham Laser Acupuncture — Sham laser acupuncture irradiation was conducted using an RJ Laser laserpen with a wavelength of 785 nm and an output power of 50 mW at the acupuncture points EXB1 and CV17, as well as BL13 and ST36 on both sides of the body. However, the laser device was not activated, and no radiation was delivered to the patient. The laser probe was positioned perpendicularly to the skin surface at the same acupuncture points, but without activating the laser. During the session, subjects wore a headset with music and protective glasses, similar to the active treatment group. The sham treatment was administered twice a week for a total of 8 sessions.
  Arms: Control Group

SUMMARY:
This clinical trial aims to evaluate the effectiveness and safety of laser acupuncture as an adjunct therapy in patients with chronic obstructive pulmonary disease (COPD). The main research questions are:

* Does laser acupuncture, when combined with standard pharmacological treatment, improve lung function (measured by FEV1% and FEV1/FVC ratio) more than sham laser acupuncture after 4 weeks of therapy?
* Does this combination also lead to better quality of life, as assessed by the COPD Assessment Test (CAT) and the St. George's Respiratory Questionnaire (SGRQ), compared to the control group, after 4 and 8 weeks?
* Is there a correlation between lung function (FEV1%) and quality of life scores (CAT and SGRQ)?
* Are there any significant adverse effects caused by laser acupuncture compared to sham treatment?

Participants will:

* Undergo spirometry and complete CAT and SGRQ questionnaires.
* Receive either laser acupuncture or sham laser acupuncture sessions.
* Return for follow-up assessments at 4 and 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with stable chronic obstructive pulmonary disease (COPD) based on the Global Initiative for COPD (GOLD).
* No acute exacerbation in the last 4 weeks.
* Male or female participants aged 20 to 80 years.
* Willing to participate in the study until completion and has signed informed consent.

Exclusion Criteria:

* History of lung surgery as treatment for COPD.
* Psychiatric or cognitive disorders.
* Underwent acupuncture within the last 2 weeks.
* Pregnant or breastfeeding.
* Presence of wounds or skin disorders at the laser acupuncture site.
* History of uncontrolled epilepsy.
* Fever > 38.0°C.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-12-10 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in One Second (FEV1%) | Baseline and 4 weeks after intervention
  Pulmonary function will be assessed using spirometry to measure the percentage of the predicted FEV1 value.
FEV1/FVC Ratio | Baseline and 4 weeks after intervention
  Pulmonary function will also be evaluated by calculating the FEV1/FVC ratio through spirometry
COPD Assessment Test (CAT) Score | Baseline, 4 weeks, and 8 weeks after intervention
  Health status and quality of life will be assessed using the CAT questionnaire, which scores from 0 to 40.
  Higher scores indicate worse health status.
St. George's Respiratory Questionnaire (SGRQ) Score | Baseline, 4 weeks, and 8 weeks after intervention
  Quality of life will be assessed using the SGRQ, which includes symptom, activity, and impact domains.
  Scores range from 0 to 100, with higher scores indicating poorer quality of life.

SECONDARY OUTCOMES:
Correlation Between FEV1% and Quality of Life Scores | Baseline, 4 weeks, and 8 weeks
  The correlation between FEV1% and CAT/SGRQ scores will be analyzed. Quality of life was assessed using the COPD Assessment Test (CAT) and the St. George's Respiratory Questionnaire (SGRQ).
  The CAT score ranges from 0 to 40, with higher scores indicating a worse impact of COPD on the patient's health status.
  The SGRQ score ranges from 0 to 100, where higher scores indicate poorer quality of life.
Adverse Events Related to Intervention | Immediately post-intervention until 8 weeks
  Any adverse events after the intervention, such as infection, pain, or skin irritation at the laser site, will be monitored and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospital
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided